CLINICAL TRIAL: NCT04499027
Title: Prognostic Value of Lung Ultrasound in Predicting Intensive Care Unit Length of Stay in Adult Cardiac Surgery: A Prospective Observational Study
Brief Title: Prognostic Value of Lung Ultrasound in Predicting Intensive Care Unit Length of Stay in Adult Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate professor of Amesthesiology, Fayoum University Hospital
Other Study IDs: D230
Record Dates: First submitted 2020-07-26; First posted 2020-08-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
Keywords: Lung ultrasound; coronary artery bypass graft (CABG); open heart surgery; ICU LOS
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound scan — 12 hours postoperatively using a convex ultrasound probe LUS will be performed by an experienced radiologist according to standardized protocols. For each hemi-thorax 3 main areas (anterior (Ant), lateral (Lt) and posterior (Post)) marked by the para-sternal, anterior axillary and posterior axillary lines will be identified. Each one will be divided into upper and lower halves, making a sum of 6 different quadrants for each side: anterior superior, anterior inferior, lateral superior, lateral inferior, posterior superior, posterior inferior.
  For each quadrant a score will be assigned based on B lines which are defined as comet like artifacts indicating subpleural interstitial edema as follows:
  (0) normal aeration: A lines with lung sliding or fewer than two isolated B lines; (1) moderate loss of lung aeration: well-defined, multiple B lines ; (2) severe loss of lung aeration: multiple coalescent B lines; and (3) complete loss of lung aeration or lung consolidation.

SUMMARY:
Being easy, bedside, non-expensive, noninvasive and radiation free, there has been a growing interest in the implementation of lung ultrasound in critical care management in the last decade, cardiac surgery was not an exception in both adult and pediatric surgeries Many predictors for open heart surgery outcomes have been studied in past years including The Society of Thoracic Surgeons (STS) risk score and the EuroSCORE (ES), preoperative clinical condition, associated chronic diseases, type of surgery, age, duration of cardiopulmonary bypass and brain natriuretic peptide (BNP), cystatin-C A recent study described the use of a novel postoperative lung ultrasound score scanning for B lines which denote subpleural interstitial edema in various lung regions for predicting critical care length of stay in pediatric cardiac surgeries.

The objective of the current study is to evaluate the role of the new lung ultrasound score in predicting the length of postoperative intensive care stay after adult open heart surgeries.

DETAILED DESCRIPTION:
After approval of the local institutional ethics committee and local institutional review board. All patients scheduled for open heart surgery in Fayoum university hospital starting from August 2020 will be enrolled in this prospective observational study until fulfilling sample size. A detailed informed consent will be signed by the eligible participants before recruitment ANESTHETIC TECHNIQUE All patients will be preoperatively assessed and investigated by complete blood count, coagulation profile, Liver and kidney functions and serum electrolytes. Chest X-ray, Electrocardiography (ECG) and echocardiography will be routinely done. Coronary angiography and carotid arterial duplex will be requested if needed.

Patient will be premedicated by 10 mg morphine intramuscularly at morning of the operation. Prior to induction of anesthesia, standard monitoring will be applied including a five-lead electrocardiography system, a pulse oximeter probe. A peripheral intravenous (IV) cannula will be placed. An arterial will be inserted using a 20 G cannula either right or left radial artery under local anesthesia. After pre-oxygenation, general anesthesia will be induced using midazolam 2-5 mg, fentanyl (3-10 μg/kg), propofol (1-1.5 mg/Kg), followed by atracurium (0.5 mg/kg).

After trachea intubation, patients will be mechanically ventilated with oxygen in air so as to achieve normocarbia. A main stream capnogram, an esophageal temperature probe and a Foley catheter will also be placed. A triple-lumen central venous catheter will be placed usually through the right internal jugular vein.

Maintenance of anesthesia will be achieved by inhaled Isoflurane 0.4 to 1% and atracurium infusion at a rate of 0.5 mg/kg/h. After initiating extracorporeal circulation, Propofol infusion at a rate of 50-100 µg/kg/min will be added to replace isoflurane inhalation.

Patients will receive intravenous heparin (300-500 IU/kg body weight) before the initiation of cardiopulmonary bypass (CPB) to achieve an activated clotting time (ACT) of more than 480 seconds. Cardiopulmonary bypass was instituted with the use of a non-pulsatile blood flow at 2.4 L/min/m2, a non-heparin-coated circuit, and a membrane oxygenator. Mean arterial pressure will be adjusted to exceed 60mmHg before, during and after cardiopulmonary bypass (CBP) . Cardiac arrest will be induced using St Thomas crystalloid solution (Hamburg). Lactated Ringer's solution will be added to the CPB circuit to maintain reservoir volume if needed, and packed red blood cells will be infused when hemoglobin level drops to less than 7g/dl. After rewarming the patient to 37°C and weaning from CPB; Protamine sulfate will be used to reverse the effect of heparin.

After skin closure and wound dressing, patients will be transferred to the intensive care unit intubated with manual ventilation and full monitoring during transfer.

Intensive care Tracheal extubation will be performed when the patient meets the following criteria: awake or arousable, hemodynamically stable, no ongoing active bleeding, warm extremities, no electrolyte abnormalities, no or minimal inotropic support and a satisfactory arterial blood gas with a fraction of inspired oxygen (FiO2) < 0.5, Ventilator pressure support reduced to 10 CmH2O with Positive End Expiratory Pressure (PEEP) 5-7 CmH2O.

ICU management and decisions will be left to the intensivist who is responsible of the postoperative cardiac critical care.

Patient will be discharged from ICU when the following criteria are met: Awake patient with oxygen saturation (SpO2) < 90% at FIO2 > 0.5 by facemask, adequate cardiac stability, no intravenous inotropic or vasopressor supportive therapy, no hemodynamically significant arrhythmia, not dependent on epicardial external pacing no major bleeding i.e. chest tube drainage less than 50 ml/h, urine output of more than 0.5 ml/kg/h and no vital threats to other organ systems such as kidneys and liver.

Lung Ultrasound scan (LUS) All patients will be examined at 12 hours postoperatively as per our institution routine using a convex ultrasound probe, any other LUS will be done upon demand.

LUS will be performed by an experienced radiologist according to standardized protocols.

This will be used to calculate total LUS-score (calculated as a sum of all quadrants score) and individual areas score.

Sample size was calculated using (G power). Minimal sample size of patients was 191 needed to get power level 0.80, alpha level 0.05 (two tailed) and 0.20 as expected β (slope of regression line) for predicting intensive care Length of stay .

Data management will be performed using the Statistical Package for Social Sciences (version 22.0; SPSS Inc., Chicago, IL, USA). Descriptive statistics (mean, standard deviation for quantitative data, and number and percentages for qualitative data) will be used to summarize the data. Nominal data will be analyzed using simple chi squared test, while independent sample t-test or one-way ANOVA procedure will be used to compare means for two or three groups of cases, respectively. Regression analysis will be performed to determine the predictors for LOS. A probability value (P value) ≤ 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* all patients Scheduled for elective cardiac surgery for valve replacement, CABG or adult congenital (VSD or ASD) via median sternotomy

Exclusion Criteria:

* subjects with inadequate acoustic windows or incomplete examinations (as defined below),
* Patients with emergency surgeries.
* Patients with thoracic deformities or preexisting pulmonary pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted in Fayoum uniersity hospital who are candidates for open heart surgeries
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Intensive care Length of stay | from ICU admission till patient discharge to ward assessed up to 30 days
  in days

SECONDARY OUTCOMES:
EURO Score II | 24 hours before operation
  calculated preoperatively using different variables which are age, gender, renal impairment, extracardiac arteriopathy, poor mobility, previous cardiac surgery, chronic lung disease, critical preoperative state, presence of insulin dependent diabetes, New York Heart Association (NYHA) classification, Canadian cardiovascular society (CCS) class, left ventricular function, recent myocardial infarction, pulmonary hypertension, urgency and weight of the operation and whether thoracic aorta is involved in surgery.18 Score will be calculated using an online calculator by QxMD website.
previous associated comorbidities | 24 hours before operation
  Diabetes, hypertension, chronic renal failure, liver impairment
primary pathology | 24 hours before operation
  Coronary artery disease, valvular heart disease
planned operative procedure | 24 hours before operation
  Coronary artery bypass graft, valve replacement, Ventricular Septal Defect repair
liver enzymes | 24 hours before operation and 1 hour after operation
  ALT
sodium level | 24 hours before operation and 1 hour after operation
  before and after the operation
potassium level | 24 hours before operation and 1 hour after operation
  before and after the operation
creatinine | 24 hours before operation and 1 hour after operation
  before and after the operation
urea | 24 hours before operation and 1 hour after operation
  before and after the operation
hemoglobin | 24 hours before operation and 1 hour after operation
  before and after the operation
platelet count | 24 hours before operation and 1 hour after operation
  before and after the operation
prothrombin concentration | 24 hours before operation and 1 hour after operation
  before and after the operation
prothrombin time | 24 hours before operation and 1 hour after operation
  before and after the operation
Cardiopulmonary Bypass (CPB) time | assessed at the end of CBP up to 12 hours from start of operation
  in minutes
Concomitant vasoactive medications | assessed at te end of the operation up to 12 hours from the start of the operation
  Noradrenaline, adrenaline, dobutamine
Arterial blood gas values | assessed up to 24 after the end of operation
  baseline after induction , before and after weaning from CBP and postoperatively in critical care with LUS
Intra and post-operative invasive BP | assessed up to 24 hours postoperatively
  (invasive BP measured in mmhg
Intra and post-operative heart rate | assessed up to 24 hours postoperatively
  Heart rate measured in beats per minute
Postoperative total LUS score | assessed 12 hours after the end of the operation
  as a sum af all areas assessed by ultrasound
individual lung areas score | assessed 12 hours after the end of the operation
  (Anterior, Lateral and Posterior).
extubation time | assessed up to 30 days
  time from ICU admission till Endotracheal tube removal
in-hospital mortality | until patient discharge assessed up to 30 days
  death before hospital discharge
Post-operative complications | assessed until patient discharge or up to 30 days postoperatively
  Myocardial infarction, atrial fibrillations, Cerebral stroke or bleeding, GI bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cantinotti M, Giordano R, Volpicelli G, Kutty S, Murzi B, Assanta N, Gargani L. Lung ultrasound in adult and paediatric cardiac surgery: is it time for routine use? Interact Cardiovasc Thorac Surg. 2016 Feb;22(2):208-15. doi: 10.1093/icvts/ivv315. Epub 2015 Nov 18. PMID 26586677
- [Background] Mojoli F, Bouhemad B, Mongodi S, Lichtenstein D. Lung Ultrasound for Critically Ill Patients. Am J Respir Crit Care Med. 2019 Mar 15;199(6):701-714. doi: 10.1164/rccm.201802-0236CI. PMID 30372119
- [Background] Bouabdallaoui N, Stevens SR, Doenst T, Petrie MC, Al-Attar N, Ali IS, Ambrosy AP, Barton AK, Cartier R, Cherniavsky A, Demondion P, Desvigne-Nickens P, Favaloro RR, Gradinac S, Heinisch P, Jain A, Jasinski M, Jouan J, Kalil RAK, Menicanti L, Michler RE, Rao V, Smith PK, Zembala M, Velazquez EJ, Al-Khalidi HR, Rouleau JL; STICH Trial Investigators. Society of Thoracic Surgeons Risk Score and EuroSCORE-2 Appropriately Assess 30-Day Postoperative Mortality in the STICH Trial and a Contemporary Cohort of Patients With Left Ventricular Dysfunction Undergoing Surgical Revascularization. Circ Heart Fail. 2018 Nov;11(11):e005531. doi: 10.1161/CIRCHEARTFAILURE.118.005531. PMID 30571194
- [Background] Wynne R. Variable definitions: implications for the prediction of pulmonary complications after adult cardiac surgery. Eur J Cardiovasc Nurs. 2004 Apr;3(1):43-52. doi: 10.1016/j.ejcnurse.2003.11.001. PMID 15053887
- [Background] Rouby JJ, Arbelot C, Gao Y, Zhang M, Lv J, An Y, Chunyao W, Bin D, Valente Barbas CS, Dexheimer Neto FL, Prior Caltabeloti F, Lima E, Cebey A, Perbet S, Constantin JM; APECHO Study Group. Training for Lung Ultrasound Score Measurement in Critically Ill Patients. Am J Respir Crit Care Med. 2018 Aug 1;198(3):398-401. doi: 10.1164/rccm.201802-0227LE. No abstract available. PMID 29557671
- See also: Euro score II — http://qxmd.com/calculate/calculator_285/euroscore-ii